CLINICAL TRIAL: NCT00451789
Title: Risk Factors of Minor Head Injury in Traumatological Patients
Brief Title: Risk Factors of Minor Head Injury
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Other Study IDs: HW1
Record Dates: First submitted 2007-03-23; First posted 2007-03-26 (Estimated); Last update posted 2007-03-26 (Estimated); Status verified 2007-03

CONDITIONS: Minor Head Injury; Intracranial Bleeding; Traumatic Brain Injury
Keywords: Minor head injury; iintracranial bleeding; traumatic brain injury; Cranial computed tomography; anticoagulatory drugs
MeSH Terms: conditions — Craniocerebral Trauma; Intracranial Hemorrhages; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Introduction and Aims:

The objective of this prospective study is to evaluate the risk factors of minor head injury in all consecutive patients of one year.

DETAILED DESCRIPTION:
Minor head injury (MHI)is one of the most common diagnoses in emergency rooms and traumatological outpatient departments. The aim of this study is to find clear evidence which risk factors are the most important in MHI patients to develop intracranial bleeding. We hypothetize that anticoagulation is one of the main risk factors for intracranial bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Minor head injury, dizziness, nausea, vomiting

Exclusion Criteria:

* no injury to the head

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12500
Dates: Start 2004-12; Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Machold, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Department for Traumatology/Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Background] Karni A, Holtzman R, Bass T, Zorman G, Carter L, Rodriguez L, Bennett-Shipman VJ, Lottenberg L. Traumatic head injury in the anticoagulated elderly patient: a lethal combination. Am Surg. 2001 Nov;67(11):1098-100. PMID 11730229
- [Background] Wojcik R, Cipolle MD, Seislove E, Wasser TE, Pasquale MD. Preinjury warfarin does not impact outcome in trauma patients. J Trauma. 2001 Dec;51(6):1147-51; discussion 1151-2. doi: 10.1097/00005373-200112000-00021. PMID 11740267
- [Derived] Wolf H, Machold W, Frantal S, Kecht M, Pajenda G, Leitgeb J, Widhalm H, Hajdu S, Sarahrudi K. Risk factors indicating the need for cranial CT scans in elderly patients with head trauma: an Austrian trial and comparison with the Canadian CT Head Rule. J Neurosurg. 2014 Feb;120(2):447-52. doi: 10.3171/2013.10.JNS13726. Epub 2013 Dec 6. PMID 24313609